CLINICAL TRIAL: NCT07137520
Title: An Observational Study on the Relationship Between Different Exercise Intensities and Energy Expenditure Metabolism
Brief Title: The Impact of Various Exercise Intensities on Energy Expenditure Metabolism
Acronym: activity
Status: Not yet recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-240615-H0893; SIATCAS (Other: Shenzhen Institutes of Advanced Technology，Chinese Academy of Sciences)
Record Dates: First submitted 2025-04-03; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Physical Activity
Keywords: Metabolic response; Energy expenditure; Physical fitness
MeSH Terms: conditions — Motor Activity | interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole blood
  * Feces
  * Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sedentary group: Godin scale score ≥ 24
  Interventions: Other: Observation without intervention
- Moderately active group: 14≥ Godin scale score ≥ 23
  Interventions: Other: Observation without intervention
- Active group: Godin scale score <14
  Interventions: Other: Observation without intervention

INTERVENTIONS:
Other: Observation without intervention — Observation without intervention

SUMMARY:
The goal of this observational study is to learn about the effects of physical activity in adult on metabolic response. The main question it aims to answer is:

* if physical activity is unlimited to increase the total energy expenditure (TEE)?

Participants will engage in the following measurements:

* Record their daily physical activity by GT3X.
* Measure TEE by doubly-labeled water (DLW) method
* Measure basal energy expenditure(BEE) and thermic effect of food(TEF) by respiratory chamber

DETAILED DESCRIPTION:
The purpose of this study is to explore the effect of various physical activities on metabolic and behavior response. Energy expenditure, body composition, and metabolism will be measured by the following measurements:

* TEE:

TEE will be measured using the DLW method. Urine samples from all participants in the DLW subset will be stored at -20℃ and shipped on dry ice for analysis in the laboratory of Prof. John Speakman at the Shenzhen Institutes of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation. TEE will then be calculated using mean CO2 production.

* REE and TEF:

REE and TEF will be measured by indirect calorimetry while participants are resting supine in a respiratory chamber with thermoneutral conditions. Oxygen consumption and CO2 production will be measured to calculate energy expenditure. REE will be consistently measured throughout sleeping at night and in the morning after overnight fasting, and TEF will be measured after breakfast.

* Physical activity：

Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day with less than 12 hours of wear. For a valid measure the goal is to get 2 weekday and 2 weekend days.

* VO2max test:

Participants need to warm up with simple stretching or light aerobic exercise before the test. The test will be conducted on a treadmill. A comfortable running speed acceptable to the participants will be set. The treadmill's incline will be increased by 10% every two minutes until the individual reaches their physical limit and can no longer continue. During this test, a respiratory mask and gas analyzer will be used to measure the concentration of oxygen (O2) and carbon dioxide (CO2) in the breath to calculate VO2max.

* Food intake

Photographic and food weighing methods to record food intake for two random days throughout the period of DLW measurement.

* Blood glucose

Fasting and post-prandial glucose will be recorded by a continuous glucose monitoring system.

* Body composition：

Fat mass will be measured by Magnetic Resonance Imaging (MRI, Shanghai united imaging, uMR 790 ).

Bioimpedance Analysis will measure fat-free mass (Tanita, MC-980). Bone mass will be measured by Dual Energy X-ray Absorptiometry (DXA, Horizon Wi, HOLOGIC).

* Body weight:

At visit 1, fasting body weight will be measured using a calibrated seca at the beginning of the visit. Fasting weight will be measured at visit 2 and, if applicable.

* Height:

Height (to +0.1 cm) will be measured by seca 217 stable without wearing shoes.

* Waist circumference:

Hip and waist circumference (to +0.3 cm) will be measured using a whole body laser scanner.

* Blood pressure:

Systolic and diastolic blood pressure will be measured using an Omron digital sphygmomanometer.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.5 kg/m2

Exclusion Criteria:

* Individuals who have undergone major surgery in the past 6 months (excluding tooth extraction);
* Individuals with severe metabolic and cardiovascular diseases such as diabetes, hypoglycemia, and hypertension;
* Individuals with exercise-related injuries, including joint diseases and fractures;
* Individuals diagnosed with infectious diseases such as HIV, tuberculosis, malaria, etc.;
* Individuals with mental and neurological disorders including anorexia nervosa;
* Individuals who have attempted weight loss or gain through various methods in the past three months;
* Individuals in preconception, pregnancy, and lactation periods;
* Individuals with autism and those with metal implants in their bodies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Shenzhen, Guangzhou, China
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Differences in total energy expenditure (TEE) measured by the doubly labeled water (DLW) method across experimental groups | 14days
  - The change in TEE will be evaluated using the DLW. Urine samples from all participants in the DLW subset will be stored at -20℃ and shipped on dry ice for analysis in the laboratory of Dr. John Speakman at the University of Aberdeen, or the Shenzhen Institutes of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation (Speakman et al 2021: Cell reports medicine). TEE will then be calculated using mean CO2 production using the Weir equation.
Differences in non-exercise physical activity across experimental groups | 14days
  - Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days.
Differences in resting energy expenditure (REE) measured by respiratory chamber across experimental groups | 1 day
  - REE will be evaluated by respiratory chamber.
Differences in thermic effect of food (TEF) measured by respiratory chamber across experimental groups | 1 day
  - TEF will be evaluated by respiratory chamber.
Differences in exercise energy expenditure (EEE) measured by COSMED across experimental groups | 1 hour
  - EEE will be evaluated using an indirect calorimetry COSMED.
Differences in food intake across experimental groups | 2 days
  Photographic and food weighing methods to record food intake for two random days throughout the period of DLW measurement

SECONDARY OUTCOMES:
Differences in sedentary time measured by GT3X accelerometer across experimental groups | 14 days
  - Sedentary time will be represented from the GT3X accelerometer.
Differences in glucose across experimental groups | 7 days
  Fasting and post-prandial glucose will be recorded by a continuous glucose monitoring system.
Differences in fat mass across experimental groups | 10 minutes
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Differences in fat-free mass across experimental groups | 2 minutes
  Fat-free mass will be measured by Bioimpedance Analysis (Tanita, MC-980).
Differences in bone mass intensity across experimental groups | 7 minutes
  Bone mass intensity will be measured by DXA( Horizon Wi, HOLOGIC)
Differences in circulating hormones across experimental groups | 1 minutes for collection, 7 days for analysis.
  The nurse will collect the fasting blood sample. Metabolomics will analyze circulating hormones and metabolites.
Differences in intestinal microbiota across experimental groups | 5 minutes for collection, 7 days for analysis.
  Feces will be collected for gut microbiome analysis of intestinal microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institutes of Advanced Technology，Chinese Academy of Sciences, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] Pontzer H, Durazo-Arvizu R, Dugas LR, Plange-Rhule J, Bovet P, Forrester TE, Lambert EV, Cooper RS, Schoeller DA, Luke A. Constrained Total Energy Expenditure and Metabolic Adaptation to Physical Activity in Adult Humans. Curr Biol. 2016 Feb 8;26(3):410-7. doi: 10.1016/j.cub.2015.12.046. Epub 2016 Jan 28. PMID 26832439
- See also: A standard calculation methodology for human doubly labeled water studies. — https://linkinghub.elsevier.com/retrieve/pii/S2666379121000148
- See also: Constrained Total Energy Expenditure and Metabolic Adaptation to Physical Activity in Adult Humans. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4803033/